CLINICAL TRIAL: NCT04029428
Title: Clinical Study of the Use of Yttrium-90 (90Y) and/or Lutecium-177 (177Lu) DOTATATE (DOTA-0-Tyr3-Octreotate) in the Treatment of Disseminated and / or Symptomatic Tumors With Somatostatin Receptor Overexpression
Brief Title: Peptide Receptor Radionuclide Therapy in the Treatment of Advanced, Non-resectable and/or Symptomatic Tumors With SSTR Overexpression
Acronym: POLNETS_PRRT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Warmia and Mazury (Other)
Collaborators: Stowarzyszenie Pacjentów i Osób Wspierających Chorych na Guzy Neuroendokrynne (Unknown)
Responsible Party: Principal Investigator, Jaroslaw B. Cwikla, MD, PhD, Professor UWM, MD, PhD, Clinical Professor; Head of Nuclear Medicine; Principal Investigator, University of Warmia and Mazury
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POLNETS_2004
Record Dates: First submitted 2019-05-19; First posted 2019-07-23 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Neuroendocrine Tumors
Keywords: PRRT - Peptide Receptor Radionuclide Therapy,; GEP-NET - Gastro-Entero-Pancreatic Neuroendocrine Tumours;; BPCs - Bronchopulmonary Carcinoids (Atypical & Typical); PPGLs - Pheochromocytomas/Paragangliomas;; NET-CUP - Neuroendocrine Tumours of unknown primary; clinical efficacy; toxcity - adverse events (AEs); OS - overall survival; PFS - progression free survival
MeSH Terms: conditions — Neuroendocrine Tumors; Paraganglioma | interventions — 90Y-octreotate, DOTA(0)-Tyr(3)-Thr(8)-; lutetium Lu 177 dotatate

STUDY DESIGN:
Intervention Model Description: Every patients from groups as follows: Gastro-Entero-Pancreatic Neuroendocrine Tumours - GEP-NET, (G1, G2 and G3), Broncho-pulmonary Carcinoids (BPCs Atypical-AC or Typical-TC), pheochromocytoma/paragangliomas (PPGLs) and neuroendocrine tumours of unknown primary (NET-CUP).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 90Y DOTATATE (Active Comparator): Therapy 90Y DOTATATE, total activity 4x3.7GBq (14.8 GBq), i.v. infusion of 90Y DOTATATE administered for 20 min. via infusion pump with co-infusion of amino-acids (AA) solution 1000ml for 1h before and then et least 6h after 90Y DOTATATE infusion. Therapy consists up to 4 cycles at 8 ± 2 weeks between each other.
  Interventions: Drug: 90Y-DOTATATE
- 177Lu DOTATATE or mix 90Y and 177Lu DOTATATE (50% each) (Experimental): Therapy 177Lu DOTATATE, total activity 4x5.55GBq (22.2 GBq), i.v. infusion of 177Lu DOTATATE administered for 20 min via infusion pump with co-infusion of amino-acids solution (AA) 1000ml for 1h before and then et least 6h after 177Lu DOTATATE infusion. Therapy consists up to 4 cycles at 8 ± 2 weeks between each other or therapy 90Y and 177Lu DOTATATE, 4x3.7GBq total activity 14.8 GBq, (mix 50% each 90Y and 177Lu), i.v. infusion of mix 90Y and 177Lu DOTATATE administered for 20 min via infusion pump with co-infusion of amino-acids (AA) solution 1000ml for 1h before and then et least 6h after 90Y and 177Lu DOTATATE infusion. Therapy consists up to 4 cycles at 8 ± 2 weeks between each other.
  Interventions: Drug: (177Lu-DOTAOTyr3)Octreotate; Drug: 90Y DOTATATE and 177Lu DOTATATE (mix each of 50%)

INTERVENTIONS:
Drug: 90Y-DOTATATE — Total activity of 90Y DOTATATE, 4x3.7GBq (14.8 GBq). Single session of i.v. infusion of 90Y DOTATATE administered for 20 min via infusion pump with co-infusion of amino-acids solution 1000ml for 1h before and then et least 6h after 90Y DOTATATE infusion. Therapy consists up to 4 cycles at 8 ± 2 weeks between each other.
  Other Names: 90Y DOTATATE
  Arms: 90Y DOTATATE
Drug: (177Lu-DOTAOTyr3)Octreotate — Total activity of 177Lu DOTATATE, 4x5.55GBq (22.2 GBq). Single session of i.v. infusion of 177Lu DOTATATE administered for 20 min via infusion pump with co-infusion of amino-acids solution 1000ml for 1h before and then et least 6h after 177Lu DOTATATE infusion. Therapy consists up to 4 cycles at 8 ± 2 weeks between each other.
  Other Names: 177Lu DOTATATE
  Arms: 177Lu DOTATATE or mix 90Y and 177Lu DOTATATE (50% each)
Drug: 90Y DOTATATE and 177Lu DOTATATE (mix each of 50%) — Total activity of 90Y DOTATATE and 177Lu DOTATATE, 4x3.7GBq (14.8 GBq 50% each 90Y and 177Lu). Single session of i.v. infusion of 90Y and 177Lu DOTATATE administered for 20 min via infusion pump with co-infusion of amino-acids solution 1000ml for 1h before and then et least 6h after 177Lu DOTATATE infusion. Therapy consists up to 4 cycles at 8 ± 2 weeks between each other.
  Other Names: 90Y DOTATATE and 177Lu DOTATATE (mix)
  Arms: 177Lu DOTATATE or mix 90Y and 177Lu DOTATATE (50% each)

SUMMARY:
This is a non-randomized phase II , open label, comparative study. Patients with advanced non-resectable and/or progressive gastro-entero-pancreatic Neuroendocrine Tumours - GEP-NET, (G1, G2 and G3), Broncho-pulmonary Carcinoids (BPCs Atypical-AC or Typical-TC), pheochromocytoma/paraganglioma (PPGLs) and neuroendocrine tumours of unknown primary (NET-CUP) with overexpression of somatostatin receptor (SSTR positive) will be enrolled in the study and will be treated using Peptide Receptor Radionuclide Therapy (PRRT) initially with Yttrium-90 (90Y) DOTATATE (DOTA-0-Tyr3-Octreotate), and then compare to Lutecium-177 (177Lu) DOTATATE or mix of both Yttrium-90 (90Y) and Lutecium-177 (177Lu) DOTATATE. Total maximum activity for Yttrium-90 up to 4x3,7GBq, for Lutecium-177 up to 4x5,55GBq (Lu-177) and for both (mix) 4x3,7GBq (90Y and 177Lu 50% each).

DETAILED DESCRIPTION:
This is a non-randomized phase II, open-label, comparative study. Patients with advanced, unresectable and/or progressive Gastro-Entero-Pancreatic Neuroendocrine Tumors - GEP-NET, (histological grade G1, G2 and G3), Broncho-Pulmonary Carcinoids (BPCs), including typical carcinoid (AC) and typical carcinoid (TC), pheochromocytoma/paragangliomas (PPGLs) and neuroendocrine tumors (cancers) of unknown primary (NET-CUP). All with overexpression of somatostatin receptor (SSTR positive) based on somatostatin receptor imaging (scintigraphy or PET), will be enrolled in this study.

Initially patients will be assigned to single arm of PRRT using yttrium-90 (90Y) DOTATATE (DOTA-0-Tyr3-Octreotate) and then patients will be non-randomly assigned to one of the two groups lutecium-177 (177Lu) DOTATATE or mix yttrium (90Y) DOTATATE and lutecium-177 (177Lu) DOTATATE (50% each). The dosages (total activity used in each group of treated patients will be as follows:

1. Total activity of 90Y DOTATATE 4x3,7GBq (14,8 GBq) for 4 cycles at 8 ± 2 weeks (400mCi)
2. Total activity of 177Lu DOTATATE 4x5,55GBq (22,2 GBq for 4 cycles at 8 ± 2 weeks (600 mCi)
3. Total activity of mix both 90Y DOTATATE and 177Lu DOTATATE (50 each) 4x3,7 GBq for 4 cycles at 8 ± 2 weeks (400mCi).

The non-randomized, phase II study design, allows for proposed initial active treatment arm using standard dose of 90Y DOTATATE and experimental treatment arm which composed of two options of PRRT with lutecium-177 DOTATATE or mix 90Y and 177Lu DOTATATE. The experimental therapy arm will be consisting of randomly allocated patients.

Subjects including in this study will be evaluated in the mixed patients' population, including GEP-NET, bronchopulmonary carcinoid (BPCs), paraganglioma/pheochromocytomas (PPGLs) and NET of unknown origin (NET-CUP).

Estimates of the original goals of the study can be assessed for each scheme separately using a two-step design using an external standard for comparison (the investigator's previous published results include standard PRRT using 90Y DOTATATE in subjects with GEP-NET).

Although the sample size in this study is not based on any specific statistical hypothesis to compare separate groups of patients those with PRRT using 90Y DOTATATE, next those with 177Lu DOTATATE and those who will receive mix 90Y and 177Lu DOTATATE.

This study design allows an objective set of clinical efficacy results in terms of PRRT responses and safety in these three treatment regimens in the same patient population, even different groups of tumors, which may be useful when planning next generation of the clinical trial using PRRT.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old, male or female, with histologically proven, well-differentiated G1/2 GEP-NET, BPCs, PPGLs or NET (cancer with unknown primary - CUP), with Ki-67 <20%, in selected cases patients with NETG3 will be included if there will be reported well/moderate morphological appearance but Ki-67>20% but less then Ki<30%; and there will be high expression of somatostatin receptor seen in functional imaging utilized functional imaging 99mTc HYNICTOC or 68Ga DOTATATE or 68Ga DOTATOC.
* The presence of high expression of somatostatin receptors demonstrated on Somatostatin Receptor Imaging using 99mTc HYNICTOC (SPECT) or 68Ga DOTATATE or 68Ga DOTATOC (PET) scans, et least as uptake in not involved liver, Krenning >2
* Non-resectable, advanced determined by an appropriately specialized surgeon or deemed not suitable for liver directed therapies where liver is the only site of disease;
* Performance status (PS) based on ECOG 0-2;
* Unresectable, advanced/metastatic progressive disease evaluated as clinical, biochemical, bad control symptoms of tumour hypersecretion or disease progression seen in imaging structural or functional.
* Adequate renal function (measured creatinine clearance > 30 ml/min by DTPA or eGFR),
* Adequate bone marrow function (Hb>8 g/d/L, WBC>2.0 x109L, ACN>1.5 x109L and PLT>80 x 103/L);
* Adequate liver function (serum total bilirubin ≤ 1.5 x ULN, and Alanine aminotransferase (ALAT), Aspartate aminotransferase (ASPAT), Alkaline phosphatase (ALP) ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver metastases)). INR ≤ 1.5 (or on a stable dose of LMW heparin for >2 weeks at time of enrollment);
* Life expectancy of at least 6 months;
* The tumor parameters that can be measured objectively as the size to be assessed in radiological studies on the basis of the RECIST 1.0;
* In the absence of the ability to measure tumor size based on RECIST criteria, they have tumor parameters that can be measured objectively as tumor markers determined in the blood or urine CgA, 5HIAA.
* Study treatment both planned and able to start within 28 days of inclusion;
* Willing and able to comply with all study requirements, including treatment, timing and/or nature of required assessments;
* Signed, written informed consent.

Exclusion Criteria:

* • Primary non-NETs;

  * Cytotoxic chemotherapy e.g. CAPTEM, or any other type of chemotherapy recorded 6 weeks before enrollment into the study;
  * Any type of biotherapy using somatostatin analogues or any targeted therapy within the last four weeks;
  * Pre-existing locoregional treatment such as radiomebolization (SIR-spheres) or HDR brachytherapy under CT control, performed in the last 6 months;
  * Major surgery/surgical therapy for any cause within two months before start of PRRT;
  * Surgical therapy of loco-regional metastases within the last three months prior to inclusion;
  * Uncontrolled metastases to the central nervous system, in the case of surgical and / or radiotherapeutic treatment, patients should remain on a stable dose of steroids for at least 2 weeks before enrollment, without deterioration of the general state associated with the presence of metastatic disease in the CNS;
  * Poorly controlled concurrent medical illness. E.g. unstable diabetes with glycosylated hemoglobin (HbA1c> 9.0), the optimal glycaemic control should be achieved before starting trial therapy);
  * Symptomatic heart failure NYHA class III or IV, congestive cardiac failure, myocardial infarction in the last 6 months, serious uncontrolled cardiac arrhythmia, unstable angina, or other serious cardiac problems;
  * Active uncontrolled infection, including Hepatitis and Hepatitis, HIV, in the case of HCV and HBV infection, the patient can be included in the study confirming the suppression of viral replication and the patient remains on the correct therapeutic dose of antiviral drugs;
  * Pregnant patients (a negative pregnancy test is required);
  * Women of childbearing age must present a negative pregnancy test at the beginning of the study and must use double barrier to contraception. Women of childbearing age are defined as menopausal if they remain menstrual for at least 1 year, or surgical sterilization or removal of the uterus before the start of the study;
  * Breast-feeding female patients;
  * Patients in a mental state who can't understand the nature, extent and possible consequences of participating in the study associated with radioisotope treatment, or there is evidence of a lack of cooperation by the patient;
  * Exclusive clinical and laboratory findings that may compromise the patient's safety or reduce the chances of obtaining satisfactory data to achieve the goal (s) of the study;
  * Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse;
  * The patient may be included in the maintenance treatment if the patient's clinical condition is stable.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2004-11-02 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
PFS - Progression Free Survival (time - months) | up to 8 years
  PFS is the time from the date of the start therapy to the date of first observation of documented disease progression or death due to any cause. Patients without tumor progression at the time of analysis will be censored at their last date of tumor evaluation.
  Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
  CT or MRI tumour assessment will be used to response evaluation. CT/MRI tumour assessment will be performed before start of PRRT and then after 6+2 weeks after last PRRT session followed by 6 months intervals during first 3 years of follow-up, after that annually. The measurement of PFS will be calculated in months.

SECONDARY OUTCOMES:
OS - Overall Survival (time months) | up to 8 years
  Overall survival is defined as the time from the date of the start therapy to the date of death due to any cause or the date of last contact (censored observation) at the date of data cut-off. The measurement of OS will be calculated in months.
Performance Status (PS) - evaluation criteria | up to 8 years
  Clinical response based on physical performance status (PS) using standard evaluation based on WHO/ECOG criteria. It will be assessed before each treatment cycle and then followed by 6 weeks after completion of therapy and then at three-month intervals. The measurement will be in the scale as follows: 0-asymptomatic, 1=symptomatic but completely ambulatory, 2=Symptomatic <50% in bed during the day, 3= Symptomatic >50% in bed during the day; 4=Bedbound; 5=Death.
Cancer Related Symptoms - assessment of clinical criteria | From date of first enrollment to the end of the follow-up, overall up to 8 years.
  Clinical response based on potential relief in the initial phase before PRRT during and after PRRT. Items will be assessed, including: appetite, malaise, pain associated with the disease, nausea, vomiting, fever, wheezing and abdominal pain or any other symptoms of advanced cancer. All of the above will be assessed as yes / no. Intensity will be recorded in the quality assessment.
  It will be evaluated before treatment, before each treatment cycle, and then 6 weeks after the end of therapy, and then at three-month intervals. The measurement will be made in the qualitative data set and categorized as improvement, stabilization or disease progression.
Hormonal overproduction symptoms - assessment of clinical criteria | From date of first enrollment to the end of the follow-up, overall up to 8 years.
  Hormonal response based on relief of symptoms of hormonal overproduction, which will be compare to clinical symptoms before PRRT, during and after PRRT during clinical follow-up. The presence of specific symptoms with hormone overproduction including: 1. Carcinoid syndrome (CS) - initial intensity of diarrhea and potential relief after PRRT (number per day), initial intensity of flushing and potential relief after PRRT (number per day). 2. Presence of heartburn in case of NET with ZES (Zollinger-Elisson syndrome) initial intensity and potential relief during PRRT and after finished PRRT during clinical follow-up. 3. Presence of hypoglycemia in case of NET with insulin overproduction (insulinoma), initial intensity of hypoglycemia before PRRT and potential relief after PRRT during clinical follow-up. The measurement will be made in a set of the qualitative data as improvement, stabilization or disease progression.
ORR - Objective Response Rate - evaluation criteria | from date of first enrollment to the end of the follow-up, overall up to 8 years.
  The evaluation of objective response will be utilized by multiphase structural imaging before and after i.v. contrast enhancement (CT or MRI). The radiological response will be based on RECIST 1.0 using standard terminology of objective response, performed before start of PRRT and then after 6+2 weeks after last PRRT therapy followed by 6 months intervals during first 3 years of follow-up, after that annually. The measurement will be made in a set of quantitative data as partial response (PR), stable disease (SD) or disease progression (DP).
Safety Assessments - Laboratory Parameters - evaluation criteria: CTCAEs ver. 4.0 | from date of first enrollment to the end of the follow-up, overall up to 8 years.
  Changes from Baseline in Hematology (WBC, RBC, platelets, haemoglobin), Blood chemistry (BUN, serum creatinine and creatinine clearance, uric acid, albumin, total bilirubin, AP, aspartate aminotransferase [AST/ASAT], alanine aminotransferase [ALT/ALAT], gamma-glutamyl transferase [γ-GT], [Na], [K], lactic dehydrogenase [LDH], glycosylated hemoglobin/hemoglobin A1c [glycoHb] and specific biomarkers Chromogranin-A (CgA) in the serum and 5-Hydroxyindoleacetic acid (5-HIAA) in the urine.
  The measurement will be made in a set of quantitative data, based on CTCAEs ver. 4.0. https://www.eortc.be/services/doc/ctc/CTCAE_4.03_2010-06-14_QuickReference_5x7.pdf
Vital Signs - heart rate - physiological parameter | from date of first enrollment to the end of the follow-up, overall up to 8 years.
  heart rate (beats per minute)
Systolic and diastolic blood pressure - physiological parameter | from date of first enrollment to the end of the follow-up, overall up to 8 years.
  mmHg.
BMI - Body Mass Index - physiological parameter | from date of first enrollment to the end of the follow-up, overall up to 8 years.
  weight (kg), height (m) Body Mass Index (BMI kg/m2). The measurement will be made in a set of quantitative data.
ECG - physiological parameter | from date of first enrollment to the end of the follow-up, overall up to 8 years.
  ECG analysis during each therapy session and clinical follow-up, including: P Wave, QRS Complex, QT Interval. The measurement will be made in a set of quantitative data.

CONTACTS AND LOCATIONS:
Locations (1):
- Centrum Diagnostyczno-Lecznicze Gammed, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caplin ME, Buscombe JR, Hilson AJ, Jones AL, Watkinson AF, Burroughs AK. Carcinoid tumour. Lancet. 1998 Sep 5;352(9130):799-805. doi: 10.1016/S0140-6736(98)02286-7. PMID 9737302
- [Background] Waldherr C, Pless M, Maecke HR, Haldemann A, Mueller-Brand J. The clinical value of [90Y-DOTA]-D-Phe1-Tyr3-octreotide (90Y-DOTATOC) in the treatment of neuroendocrine tumours: a clinical phase II study. Ann Oncol. 2001 Jul;12(7):941-5. doi: 10.1023/a:1011160913619. PMID 11521799
- [Background] Paganelli G, Zoboli S, Cremonesi M, Bodei L, Ferrari M, Grana C, Bartolomei M, Orsi F, De Cicco C, Macke HR, Chinol M, de Braud F. Receptor-mediated radiotherapy with 90Y-DOTA-D-Phe1-Tyr3-octreotide. Eur J Nucl Med. 2001 Apr;28(4):426-34. doi: 10.1007/s002590100490. PMID 11357492
- [Background] Reubi JC, Schar JC, Waser B, Wenger S, Heppeler A, Schmitt JS, Macke HR. Affinity profiles for human somatostatin receptor subtypes SST1-SST5 of somatostatin radiotracers selected for scintigraphic and radiotherapeutic use. Eur J Nucl Med. 2000 Mar;27(3):273-82. doi: 10.1007/s002590050034. PMID 10774879
- [Background] Kwekkeboom DJ, Bakker WH, Kam BL, Teunissen JJ, Kooij PP, de Herder WW, Feelders RA, van Eijck CH, de Jong M, Srinivasan A, Erion JL, Krenning EP. Treatment of patients with gastro-entero-pancreatic (GEP) tumours with the novel radiolabelled somatostatin analogue [177Lu-DOTA(0),Tyr3]octreotate. Eur J Nucl Med Mol Imaging. 2003 Mar;30(3):417-22. doi: 10.1007/s00259-002-1050-8. Epub 2003 Jan 9. PMID 12634971
- [Background] Esser JP, Krenning EP, Teunissen JJ, Kooij PP, van Gameren AL, Bakker WH, Kwekkeboom DJ. Comparison of [(177)Lu-DOTA(0),Tyr(3)]octreotate and [(177)Lu-DOTA(0),Tyr(3)]octreotide: which peptide is preferable for PRRT? Eur J Nucl Med Mol Imaging. 2006 Nov;33(11):1346-51. doi: 10.1007/s00259-006-0172-9. Epub 2006 Jul 18. PMID 16847654
- [Background] Waldherr C, Pless M, Maecke HR, Schumacher T, Crazzolara A, Nitzsche EU, Haldemann A, Mueller-Brand J. Tumor response and clinical benefit in neuroendocrine tumors after 7.4 GBq (90)Y-DOTATOC. J Nucl Med. 2002 May;43(5):610-6. PMID 11994522
- [Background] Cwikla JB, Sankowski A, Seklecka N, Buscombe JR, Nasierowska-Guttmejer A, Jeziorski KG, Mikolajczak R, Pawlak D, Stepien K, Walecki J. Efficacy of radionuclide treatment DOTATATE Y-90 in patients with progressive metastatic gastroenteropancreatic neuroendocrine carcinomas (GEP-NETs): a phase II study. Ann Oncol. 2010 Apr;21(4):787-794. doi: 10.1093/annonc/mdp372. Epub 2009 Oct 15. PMID 19833821
- [Background] Chinol M, Bodei L, Cremonesi M, Paganelli G. Receptor-mediated radiotherapy with Y-DOTA-DPhe-Tyr-octreotide: the experience of the European Institute of Oncology Group. Semin Nucl Med. 2002 Apr;32(2):141-7. doi: 10.1053/snuc.2002.31563. PMID 11965609
- [Background] Kwekkeboom DJ, de Herder WW, Kam BL, van Eijck CH, van Essen M, Kooij PP, Feelders RA, van Aken MO, Krenning EP. Treatment with the radiolabeled somatostatin analog [177 Lu-DOTA 0,Tyr3]octreotate: toxicity, efficacy, and survival. J Clin Oncol. 2008 May 1;26(13):2124-30. doi: 10.1200/JCO.2007.15.2553. PMID 18445841
- [Background] Bushnell DL Jr, O'Dorisio TM, O'Dorisio MS, Menda Y, Hicks RJ, Van Cutsem E, Baulieu JL, Borson-Chazot F, Anthony L, Benson AB, Oberg K, Grossman AB, Connolly M, Bouterfa H, Li Y, Kacena KA, LaFrance N, Pauwels SA. 90Y-edotreotide for metastatic carcinoid refractory to octreotide. J Clin Oncol. 2010 Apr 1;28(10):1652-9. doi: 10.1200/JCO.2009.22.8585. Epub 2010 Mar 1. PMID 20194865